CLINICAL TRIAL: NCT04171401
Title: Maximum Weight-shifts in Sitting in Non-ambulatory People With Stroke Are Related With Trunk Control and Balance in Sitting and Standing
Brief Title: Limits of Stability in Sitting in Healthy Controls and Participants Post Stroke
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Evelien Wiskerke, Physiotherapist and Researcher, MSc, PhD Candidate, KU Leuven
Other Study IDs: S57757
Record Dates: First submitted 2019-11-18; First posted 2019-11-20 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Stroke; Balance; Distorted
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Participants post stroke: Severly affected patients in the subacute phase post stroke that are unable to walk without the help of one or two therapists to assist for balance and weight-carrying. Participants were able to sit independently for two minutes. Participants post stroke performed limits of stability testing in sitting, and tests for trunk control and functional balance.
  Interventions: Other: In-patient stroke rehabilitation.
- Healthy controls: Healthy control subjects who matched patients post stroke for age and gender, and had no limitations to perform measurements. Healthy controls performed limits of stability measurements and a clinical measurements for balance.

INTERVENTIONS:
Other: In-patient stroke rehabilitation. — An in-patient multi-disciplinary stroke rehabilitation program was performed.
  Groups: Participants post stroke

SUMMARY:
In this cross-sectional study we will compare the limits of stability in non-ambulatory participants post stroke compared to healthy controls. This will be done by placing participants in a seated position on a force platform, that will measure centre of pressure displacements during a leaning task in multiple directions. The results of the limits of stability test will be compared to standard clinical Measures of trunk control and functional balance, to see if there is a relationship between both ways of measuring. And how balance and trunk control are affected in the subacute stroke population.

ELIGIBILITY:
Inclusion Criteria Participants post Stroke:

* a stroke with clear hemiplegia (a previous stroke is accepted when complete recovery was achieved)
* being a patient at the UZ Pellenberg
* Functional Ambulation Catergory of two or less
* to be able to sit independently for 2 minutes
* to be cooperative enough to fulfill multiple Evaluations and tests
* to be able to understand simple instructions and be able to execute those.

Exclusion Criteria Participants post Stroke:

* to have musculoskeletal and/or other neurological disorders that could influence the protocol
* severe communication, memory or language disorders that could disturb the understanding of the research protocol.
* no signed informed consent

Inclusion criteria healthy controls:

* Age above 50
* to be able to stand independently for 2 minutes

Exclusion criteria healthy controls:

* a disorder that could influence balance capabilities
* Berg Balance Scale less than 50 Points
* no signed informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of patients post stroke which are severly affected and are unable to walk without help of one or two persons who help cary their weight or control their balance. Participants are in the subacute phase post stroke and are admitted to a rehabilitation programme at the UZ Pellenberg.
  Healthy controls were also included in this study.
Sampling Method: Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2015-05-11 (Actual); Primary Completion 2016-01-27 (Actual); Study Completion 2016-01-27 (Actual)

PRIMARY OUTCOMES:
Limits of Stability Testing | Baseline
  The centre of pressure(COP) movement is measured while the patient is seated on a force platform and is asked by the software that is projected on a screen, to lean with the trunk in a certain direction and hold this position before going back to the starting position. The COP distance between start and end position is calculated, as well as the COP length of the trajectory that it takes the participant to reach his or her maximum leaning position.
Berg Balance Scale | Baseline
  The Berg Balance Scale (BBS) is used to assess functional balance. The scale consists of 14 items, for each item the minimum score is 0 points, the maximum score is 4 points. A total amount of 56 points can be achieved on the Berg Balance Scale which indicates a normal balance for adults. A score lower than 45 points in elderly indicates that individuals may be at greater risk of falling.
Trunk Impairment Scale | Baseline
  The Trunk Impairment Scale (TIS) assesses static and dynamic sitting balance and coordination of trunk movement. The test consists of 17 items with a minimum score of 0 and a maximum score of 23 points, which is calculated by adding up the scores from the subscales (0-7 Points for static sitting Balance, 0-10 Points for dynamic sitting Balance, 0-6 Points for coordination), with a higher scores for better trunk control.
Trunk Control Test | Baseline
  The Trunk Control Tests consists of four items with a maximum score of 100 points. The patient is asked to turn in bed, come from lying to sitting at the bedside and stay seated at the bedside. A higher score shows better functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Geert Verheyden, Study Director — KU Leuven